CLINICAL TRIAL: NCT01088503
Title: The TRANSLATE-ACS Study: Treatment With ADP Receptor Inhibitors: Longitudinal Assessment of Treatment Patterns and Events After Acute Coronary Syndrome
Brief Title: Treatment With Adenosine Diphosphate (ADP) Receptor Inhibitors: Longitudinal Assessment of Treatment Patterns and Events After Acute Coronary Syndrome
Acronym: TRANSLATE-ACS
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: 12549; H7T-US-B007 (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ADP receptor inhibitor treatment: Participants admitted for non ST elevation myocardial infarction (NSTEMI) or ST elevation myocardial infarction (STEMI) undergoing percutaneous coronary intervention (PCI) and treated with an ADP receptor inhibitor during the index hospitalization.
  Interventions: Drug: ADP receptor inhibitors

INTERVENTIONS:
Drug: ADP receptor inhibitors — Dosage regimen as determined by the treating physician.

SUMMARY:
The TReatment with ADP receptor iNhibitorS: Longitudinal Assessment of Treatment Patterns and Events after Acute Coronary Syndrome (TRANSLATE-ACS) study is a prospective, observational longitudinal study to evaluate the real world effectiveness and use of prasugrel and other ADP receptor inhibitor therapies among myocardial infarction (MI) participants treated with percutaneous coronary intervention (PCI) during the index hospitalization. Participant management and treatment decisions are at the discretion of the care team per routine clinical practice. Approximately 17,000 participants will be enrolled at approximately 350 sites in the United States. Follow-up will be conducted through 15 months in approximately 15,650 participants.

TRANSLATE-ACS will complement the results of both randomized controlled clinical trials and current registries in addressing the real world treatment patterns and clinical outcomes for MI participants managed with PCI and initiated on ADP receptor inhibitor therapy. In addition to determining the effectiveness of prasugrel in comparison to other ADP receptor inhibitors, the study will also determine factors associated with initial ADP receptor inhibitor selection and longitudinal patterns of use, evaluate the safety, and describe and compare resource use and medical costs associated with ADP receptor inhibitors. Additionally, this study will generate a continuum of information from the inpatient to outpatient settings to provide a comprehensive picture of participant treatment and outcomes not currently available for novel ADP receptor inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age
* diagnosed with NSTEMI or STEMI treated with a PCI during the index hospitalization
* initiated (or continued) on ADP receptor inhibitor therapy before discharge
* fully informed and are able to provide written consent for longitudinal follow-up and data collection

Exclusion Criteria:

* simultaneously participating in a research study that directs choice of either an investigational or approved ADP receptor inhibitor within the first 12 months after MI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants admitted or already in hospital with acute myocardial infarction (MI) who are treated with percutaneous coronary intervention (PCI) and an ADP receptor inhibitor.
Sampling Method: Non-Probability Sample
Enrollment: 12227 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours EST), Study Director — Eli Lilly and Company
Locations (186):
- United States (185):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anchorage, Alaska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fayetteville, Alaska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gilbert, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Smith, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rogers, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berkeley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Loma Linda, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roseville, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salinas, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Barbara, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockton, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thousand Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parker, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bridgeport, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Farmington, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hartford, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newark, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlantis, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brandon, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hudson, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakeland, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stuart, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vero Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellington, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winter Haven, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riverdale, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carbondale, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Geneva, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoffman Estates, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Joliet, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oak Lawn, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rock Island, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockford, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Urbana, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elkhart, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Wayne, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hammond, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Muncie, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Davenport, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Overland Park, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Crestview Hills, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Owensboro, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alexandria, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewiston, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Annapolis, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cumberland, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hagerstown, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salisbury, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takoma Park, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bay City, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dearborn, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flint, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Blanc, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marquette, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Clemens, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saginaw, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Joseph, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southfield, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warren, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wyoming, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coon Rapids, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duluth, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edina, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Cloud, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Joplin, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bozeman, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalispell, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bridgewater, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherry Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Brunswick, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newark, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ridgewood, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Summit, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elmira, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnson City, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stony Brook, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Utica, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valhalla, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lumberton, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Canton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kettering, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleburg Heights, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Youngstown, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bend, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tualatin, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Abington, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allentown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bryn Mawr, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camp Hill, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Darby, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensburg, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harrisburg, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hershey, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnstown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Langhorne, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sayre, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uniontown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anderson, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grapevine, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Round Rock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Temple, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesapeake, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport News, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roanoke, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Virginia Beach, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winchester, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Everett, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntington, West Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Green Bay, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Racine, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waukesha, Wisconsin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras, Puerto Rico

REFERENCES:
- [Derived] Rymer JA, Kaltenbach LA, Doll JA, Messenger JC, Peterson ED, Wang TY. Safety of Dual-Antiplatelet Therapy After Myocardial Infarction Among Patients With Chronic Kidney Disease. J Am Heart Assoc. 2019 May 21;8(10):e012236. doi: 10.1161/JAHA.119.012236. PMID 31070112
- [Derived] Warraich HJ, Kaltenbach LA, Fonarow GC, Peterson ED, Wang TY. Adverse Change in Employment Status After Acute Myocardial Infarction: Analysis From the TRANSLATE-ACS Study. Circ Cardiovasc Qual Outcomes. 2018 Jun;11(6):e004528. doi: 10.1161/CIRCOUTCOMES.117.004528. PMID 29895612
- [Derived] Fanaroff AC, Kaltenbach LA, Peterson ED, Akhter MW, Effron MB, Henry TD, Wang TY. Antiplatelet Therapy Changes for Patients With Myocardial Infarction With Recurrent Ischemic Events: Insights Into Contemporary Practice From the TRANSLATE-ACS (Treatment With ADP Receptor Inhibitors: Longitudinal Assessment of Treatment Patterns and Events After Acute Coronary Syndrome) Study. J Am Heart Assoc. 2018 Feb 8;7(4):e007982. doi: 10.1161/JAHA.117.007982. PMID 29437596
- [Derived] Tisminetzky M, Wang TY, Gurwitz J, Kaltenbach LA, McManus D, Gore J, Peterson E, Goldberg RJ. Magnitude and Characteristics of Patients Who Survived an Acute Myocardial Infarction. J Am Heart Assoc. 2017 Sep 25;6(9):e006373. doi: 10.1161/JAHA.117.006373. PMID 28947562
- [Derived] Guimaraes PO, Krishnamoorthy A, Kaltenbach LA, Anstrom KJ, Effron MB, Mark DB, McCollam PL, Davidson-Ray L, Peterson ED, Wang TY. Accuracy of Medical Claims for Identifying Cardiovascular and Bleeding Events After Myocardial Infarction : A Secondary Analysis of the TRANSLATE-ACS Study. JAMA Cardiol. 2017 Jul 1;2(7):750-757. doi: 10.1001/jamacardio.2017.1460. PMID 28538984
- [Derived] Hess CN, Kaltenbach LA, Doll JA, Cohen DJ, Peterson ED, Wang TY. Race and Sex Differences in Post-Myocardial Infarction Angina Frequency and Risk of 1-Year Unplanned Rehospitalization. Circulation. 2017 Feb 7;135(6):532-543. doi: 10.1161/CIRCULATIONAHA.116.024406. PMID 28153990
- [Derived] Jackson LR 2nd, Peterson ED, McCoy LA, Ju C, Zettler M, Baker BA, Messenger JC, Faries DE, Effron MB, Cohen DJ, Wang TY. Impact of Proton Pump Inhibitor Use on the Comparative Effectiveness and Safety of Prasugrel Versus Clopidogrel: Insights From the Treatment With Adenosine Diphosphate Receptor Inhibitors: Longitudinal Assessment of Treatment Patterns and Events After Acute Coronary Syndrome (TRANSLATE-ACS) Study. J Am Heart Assoc. 2016 Oct 21;5(10):e003824. doi: 10.1161/JAHA.116.003824. PMID 27792656
- [Derived] Fosbol EL, Ju C, Anstrom KJ, Zettler ME, Messenger JC, Waksman R, Effron MB, Baker BA, Cohen DJ, Peterson ED, Wang TY. Early Cessation of Adenosine Diphosphate Receptor Inhibitors Among Acute Myocardial Infarction Patients Treated With Percutaneous Coronary Intervention: Insights From the TRANSLATE-ACS Study (Treatment With Adenosine Diphosphate Receptor Inhibitors: Longitudinal Assessment of Treatment Patterns and Events After Acute Coronary Syndrome). Circ Cardiovasc Interv. 2016 Nov;9(11):e003602. doi: 10.1161/CIRCINTERVENTIONS.115.003602. PMID 27789517
- [Derived] Krishnamoorthy A, Peterson ED, Knight JD, Anstrom KJ, Effron MB, Zettler ME, Davidson-Ray L, Baker BA, McCollam PL, Mark DB, Wang TY. How Reliable are Patient-Reported Rehospitalizations? Implications for the Design of Future Practical Clinical Studies. J Am Heart Assoc. 2016 Jan 25;5(1):e002695. doi: 10.1161/JAHA.115.002695. PMID 26811163
- [Derived] Hess CN, Wang TY, McCoy LA, Messenger JC, Effron MB, Zettler ME, Henry TD, Peterson ED, Fonarow GC. Unplanned Inpatient and Observation Rehospitalizations After Acute Myocardial Infarction: Insights From the Treatment With Adenosine Diphosphate Receptor Inhibitors: Longitudinal Assessment of Treatment Patterns and Events After Acute Coronary Syndrome (TRANSLATE-ACS) Study. Circulation. 2016 Feb 2;133(5):493-501. doi: 10.1161/CIRCULATIONAHA.115.017001. Epub 2015 Dec 17. PMID 26680241
- [Derived] Wang TY, Henry TD, McCoy LA, Berger PB, Cohen DJ, Effron MB, Zettler M, Baker BA, Messenger JC, Peterson ED. Contemporary use of platelet function and pharmacogenomic testing among patients with acute myocardial infarction undergoing percutaneous coronary intervention in the United States. Am Heart J. 2015 Oct;170(4):706-14. doi: 10.1016/j.ahj.2015.06.021. Epub 2015 Jul 2. PMID 26386794
- [Derived] Mathews R, Wang TY, Honeycutt E, Henry TD, Zettler M, Chang M, Fonarow GC, Peterson ED; TRANSLATE-ACS Study Investigators. Persistence with secondary prevention medications after acute myocardial infarction: Insights from the TRANSLATE-ACS study. Am Heart J. 2015 Jul;170(1):62-9. doi: 10.1016/j.ahj.2015.03.019. Epub 2015 Apr 2. PMID 26093865
- [Derived] Mathews R, Peterson ED, Honeycutt E, Chin CT, Effron MB, Zettler M, Fonarow GC, Henry TD, Wang TY. Early Medication Nonadherence After Acute Myocardial Infarction: Insights into Actionable Opportunities From the TReatment with ADP receptor iNhibitorS: Longitudinal Assessment of Treatment Patterns and Events after Acute Coronary Syndrome (TRANSLATE-ACS) Study. Circ Cardiovasc Qual Outcomes. 2015 Jul;8(4):347-56. doi: 10.1161/CIRCOUTCOMES.114.001223. Epub 2015 Jun 2. PMID 26038524
- [Derived] Wang TY, Henry TD, Effron MB, Honeycutt E, Hess CN, Zettler ME, Cohen DJ, Baker BA, Berger PB, Anstrom KJ, Angiolillo DJ, Peterson ED; TRANSLATE-POPS Investigators. Cluster-randomized clinical trial examining the impact of platelet function testing on practice: the treatment with adenosine diphosphate receptor inhibitors: longitudinal assessment of treatment patterns and events after acute coronary syndrome prospective open label antiplatelet therapy study. Circ Cardiovasc Interv. 2015 Jun;8(6):e001712. doi: 10.1161/CIRCINTERVENTIONS.114.001712. PMID 26025216
- [Derived] Xian Y, Wang TY, McCoy LA, Effron MB, Henry TD, Bach RG, Zettler ME, Baker BA, Fonarow GC, Peterson ED. Association of Discharge Aspirin Dose With Outcomes After Acute Myocardial Infarction: Insights From the Treatment with ADP Receptor Inhibitors: Longitudinal Assessment of Treatment Patterns and Events after Acute Coronary Syndrome (TRANSLATE-ACS) Study. Circulation. 2015 Jul 21;132(3):174-81. doi: 10.1161/CIRCULATIONAHA.114.014992. Epub 2015 May 20. PMID 25995313
- [Derived] Bagai A, Peterson ED, Honeycutt E, Effron MB, Cohen DJ, Goodman SG, Anstrom KJ, Gupta A, Messenger JC, Wang TY. In-hospital switching between adenosine diphosphate receptor inhibitors in patients with acute myocardial infarction treated with percutaneous coronary intervention: Insights into contemporary practice from the TRANSLATE-ACS study. Eur Heart J Acute Cardiovasc Care. 2015 Dec;4(6):499-508. doi: 10.1177/2048872614564082. Epub 2014 Dec 16. PMID 25515725
- [Derived] Hess CN, McCoy LA, Duggirala HJ, Tavris DR, O'Callaghan K, Douglas PS, Peterson ED, Wang TY. Sex-based differences in outcomes after percutaneous coronary intervention for acute myocardial infarction: a report from TRANSLATE-ACS. J Am Heart Assoc. 2014 Feb 7;3(1):e000523. doi: 10.1161/JAHA.113.000523. PMID 24510115
- [Derived] Wang TY, McCoy L, Henry TD, Effron MB, Messenger JC, Cohen DJ, Mark DB, Stone GW, Zettler M, Singh M, Fonarow GC, Peterson ED; TRANSLATE-ACS Study Investigators. Early post-discharge bleeding and antiplatelet therapy discontinuation among acute myocardial infarction patients treated with percutaneous coronary intervention. J Am Coll Cardiol. 2014 Apr 29;63(16):1700-2. doi: 10.1016/j.jacc.2013.12.012. Epub 2014 Jan 30. No abstract available. PMID 24486275
- [Derived] Chin CT, Wang TY, Anstrom KJ, Zhu B, Maa JF, Messenger JC, Ryan KA, Davidson-Ray L, Zettler M, Effron MB, Mark DB, Peterson ED. Treatment with adenosine diphosphate receptor inhibitors-longitudinal assessment of treatment patterns and events after acute coronary syndrome (TRANSLATE-ACS) study design: expanding the paradigm of longitudinal observational research. Am Heart J. 2011 Nov;162(5):844-51. doi: 10.1016/j.ahj.2011.08.021. PMID 22093200

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Centralized follow-up visits were conducted for all participants. Participants who completed 15-month active follow-up were considered to have completed the study.
Groups:
- Prasugrel: Participants who were admitted for non ST elevation myocardial infarction (NSTEMI) or ST elevation myocardial infarction (STEMI) underwent percutaneous coronary intervention (PCI) and were treated with prasugrel during the index hospitalization. Dosage regimen was determined by the treating physician.
- Clopidogrel: Participants who were admitted for NSTEMI or STEMI underwent PCI and were treated with clopidogrel during the index hospitalization. Dosage regimen was determined by the treating physician.
- Ticlopidine/Ticagrelor: Participants who were admitted for NSTEMI or STEMI underwent PCI and were treated with ticlopidine or ticagrelor during the index hospitalization. Dosage regimen was determined by the treating physician.
Period: Overall Study
Arm/Group | Prasugrel | Clopidogrel | Ticlopidine/Ticagrelor
Started | 3123 | 8846 | 258
Completed | 2941 | 8161 | 241
Not Completed | 182 | 685 | 17
Not completed — Withdrawal by Subject | 118 | 327 | 10
Not completed — Death | 64 | 358 | 7

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Prasugrel: Participants who were admitted for NSTEMI or STEMI underwent PCI and were treated with prasugrel during the index hospitalization. Dosage regimen was determined by the treating physician.
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Clopidogrel | Ticlopidine/Ticagrelor | Total
Number analyzed (Participants) | 3123 | 8846 | 258 | 12227
Age, Customized [Number; unit: participants]
  ≥75 years | 88 | 1341 | 33 | 1462
  <75 years | 3035 | 7505 | 225 | 10765
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 672 | 2671 | 91 | 3434
  Male | 2451 | 6175 | 167 | 8793
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 129 | 271 | 13 | 413
  Not Hispanic or Latino | 2986 | 8525 | 244 | 11755
  Unknown or Not Reported | 8 | 50 | 1 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 35 | 39 | 0 | 74
  Asian | 55 | 94 | 1 | 150
  Native Hawaiian or Other Pacific Islander | 12 | 13 | 0 | 25
  Black or African American | 237 | 820 | 30 | 1087
  White | 2750 | 7778 | 225 | 10753
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 34 | 102 | 2 | 138
Region of Enrollment [Number; unit: participants]
  United States | 3123 | 8846 | 258 | 12227

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Adverse Cardiovascular Events (MACE)
Description: MACE is defined as a composite of all-cause death, myocardial infarction (MI), stroke, or unplanned coronary revascularization. Events that occurred more than 7 days after medication was switched or discontinued were excluded from the analysis. Observed (unadjusted) percentages of participants with MACE, as well as the statistical analyses adjusted for baseline cohort differences, are presented. Percentage of participants = (number of participants with events in 12 months/ number of participants treated) * 100.
Time Frame: Baseline through 12 months
Population: Participants who were treated with prasugrel or clopidogrel. Participants with MACE events dated prior to index PCI were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 3123 | 8838
percentage of participants | 13.14 [11.79 to 14.48] | 17.12 [16.25 to 17.98]
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.7108, Log Rank — Statistical analysis adjusted for the differences in baseline characteristics between participants treated with prasugrel vs. clopidogrel using propensity scoring; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.88 to 1.22]

2. Primary Outcome: Factors Associated With Initial Adenosine Diphosphate (ADP) Receptor Inhibitor Selection at Enrollment
Description: Factors are drug-eluting stent (DES) vs. bare metal stent (BMS) placement, other (no stent) vs. BMS, STEMI, other race, cardiogenic shock occurred within 24 hours, male, European Quality of Life Questionnaire-5 Dimension Health State Score (EQ-5D) - United States (US) Index =1 vs. <1, married, diabetes, and other vs. BMS placement. The EQ-5D US index is a participant-rated, health-related, quality-of-life instrument based on US population. Scores range from -0.11 to 1.0 with 1.0 = perfect health.
Time Frame: Day 0 (study enrollment)
Population: All enrolled participants
Measure: Number; unit: participants
Groups:
- Other: Participants who were admitted for NSTEMI or STEMI underwent PCI and were treated with clopidogrel, or ticlopidine, or ticagrelor during the index hospitalization. Dosage regimen was determined by the treating physician
Arm/Group | Prasugrel | Other
Number analyzed (Participants) | 3123 | 9104
participants
  Received DES | 2365 | 6282
  Received only BMS | 672 | 2491
  STEMI | 1831 | 4508
  Other Race (Non-Caucasian) | 365 | 1049
  Cardiogenic Shock on Presentation | 79 | 176
  Male Participants | 2451 | 6342
  EQ-5D US index = 1 vs. <1 | 1516 | 3873
  Married Participants | 2044 | 5601
  Participant has Diabetes | 767 | 2472
  No BMS or DES | 86 | 331
Statistical Analysis 1: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio (OR) = 1.464 — Odds Ratio for selection of Prasugrel for participants with DES vs BMS
Statistical Analysis 2: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio (OR) = 1.230 — Odds Ratio for selection of Prasugrel for participants with STEMI vs not STEMI
Statistical Analysis 3: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio, log = 1.657 — Odds Ratio for selection of Prasugrel for participants who were Other Race vs Caucasian
Statistical Analysis 4: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio, log = 1.684 — Odds Ratio for selection of Prasugrel for participants who had cardiogenic shock within 24 hours vs no cardiogenic shock within 24 hours
Statistical Analysis 5: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio (OR) = 1.195 — Odds Ratio for selection of Prasugrel for participants who were male vs not male
Statistical Analysis 6: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio (OR) = 1.120 — Odds Ratio for selection of Prasugrel for participants with EQ-5D US index = 1 vs. <1
Statistical Analysis 7: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio (OR) = 1.116 — Odds Ratio for selection of Prasugrel for participants who were married vs not married
Statistical Analysis 8: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio (OR) = 1.125 — Odds Ratio for selection of Prasugrel for participants who had diabetes vs no diabetes
Statistical Analysis 9: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio (OR) = 1.172 — Odds Ratio for selection of Prasugrel for participants with no BMS or DES placement vs BMS

3. Secondary Outcome: Percentage of Participants With Cumulative Severe or Moderate Bleeding Events
Description: Bleeding events were collected utilizing the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries (GUSTO) definition of bleeding. Non-coronary artery bypass grafting (CABG)-related GUSTO severe or life-threatening bleeding is any intracranial hemorrhage (ICH) OR any bleeding event resulting in substantial hemodynamic compromise requiring treatment. Non-CABG-related GUSTO moderate bleeding is any bleeding event resulting in the need for transfusion that is not considered a GUSTO severe or life-threatening bleed. Additional bleeding events are fatal bleeding or ICH, or any non -fatal surgical-related bleeding events leading to ≥4 units of red cell transfusion. Observed (unadjusted) percentages of participants with bleeding events, as well as the statistical analyses adjusted for baseline cohort differences, are presented. Percentage of participants = (number of participants with events / number of participants treated) * 100.
Time Frame: Baseline, 1, 6, 12 and 15 months
Population: Participants who were treated with prasugrel or clopidogrel. Participants with bleeding events dated prior to index PCI were excluded from the analysis. The analysis was based on the initial treatment assignment, regardless of whether or not the participants switched or discontinued that treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 3123 | 8833
percentage of participants
  Baseline | 0.54 [0.34 to 0.87] | 0.45 [0.33 to 0.62]
  1 month | 1.22 [0.89 to 1.67] | 1.62 [1.38 to 1.91]
  6 months | 1.93 [1.50 to 2.48] | 2.77 [2.45 to 3.13]
  12 months | 2.72 [2.20 to 3.36] | 3.86 [3.48 to 4.29]
  15 months | 3.10 [2.55 to 3.79] | 4.21 [3.81 to 4.66]
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.1882, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.88 to 1.93] — Hazard ratio (HR) is for the analysis at 12 months

4. Secondary Outcome: Percentage of Participants With MACE and Who Had No Prior History of Transient Ischemic Attack (TIA)/Stroke, Weigh ≥60 Kilograms (kg), and Are Age <75 Years
Description: MACE is defined as a composite of all-cause death, MI, stroke, or unplanned coronary revascularization. Events that occurred more than 7 days after medication was switched or discontinued were excluded from the analysis. Observed (unadjusted) percentages of participants with MACE, as well as the statistical analyses adjusted for baseline cohort differences, are presented. Percentage of participant = (number of participants with events / number of participants treated) * 100.
Time Frame: Baseline through 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 3123 | 8838
percentage of participants | 12.67 [11.3 to 14.03] | 15.89 [14.92 to 16.85]
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; Hazard Ratio (HR) = 0.967, 95% CI 2-sided [0.849 to 1.103] — Statistical analysis adjusted for the differences in baseline characteristics between participants treated with prasugrel vs. clopidogrel using propensity scoring

5. Secondary Outcome: Percentage of Participants With MACE Over 1, 6 and 15 Months
Description: MACE is defined as a composite of all-cause death, MI, stroke, or unplanned coronary revascularization. Events that occurred more than 7 days after medication was switched or discontinued were excluded from the analysis. Observed (unadjusted) percentages of participants with MACE are presented. Kaplan-Meier analysis was used to estimate the percentage of participants with a MACE event.
Time Frame: Baseline through 1, 6 and 15 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 3123 | 8838
percentage of participants
  1 month | 4.63 [3.87 to 5.39] | 5.40 [4.88 to 5.85]
  6 months | 9.64 [8.50 to 10.77] | 12.04 [11.31 to 12.77]
  15 months | 14.26 [12.82 to 15.70] | 19.13 [18.20 to 20.07]

6. Secondary Outcome: Percentage of Participants With Definite or Probable Stent Thrombosis (ST) Events
Description: Academic Research Consortium (ARC) criteria were used to define ST. Definite ST is angiographic or pathologic confirmation of partial or total thrombotic occlusion within the peri-stent region, and at least 1 of the following additional criteria: acute ischemic symptoms; ischemic electrocardiogram changes; elevated cardiac biomarkers. Probable ST is any unexplained death within 30 days of stent implantation; any MI, which is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of ST and in the absence of any other obvious cause. Events that occurred more than 7 days after medication was switched or discontinued were excluded from the analysis. Observed (unadjusted) percentages of participants with ST events are presented. Kaplan-Meier analysis was used to estimate the percentage of participants with a definite or probable ST event.
Time Frame: Baseline through 15 months
Population: Participants who were treated with prasugrel or clopidogrel.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 3123 | 8846
percentage of participants | 1.35 [0.85 to 1.85] | 1.79 [1.49 to 2.10]

7. Secondary Outcome: Resource Use Patterns, Cumulative Total Medical Costs, and Cost Effectiveness
Time Frame: 15 months
Population: Zero participants were analyzed. Exploratory analysis of resource use patterns, cumulative total medical costs, and cost effectiveness was dependent on effectiveness in the primary outcome. As there was no effectiveness on the primary outcome demonstrated, no analysis of these outcome measure was conducted.
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Factors Associated With Initial ADP Receptor Inhibitor Selection at Enrollment: Pre-Procedure Hemoglobin
Time Frame: Day 0 (study enrollment)
Population: All enrolled participants who had pre-procedure hemoglobin evaluation.
Measure: Mean (Standard Deviation); unit: grams/deciliter (g/dL)
Arm/Group | Prasugrel | Other
Number analyzed (Participants) | 2806 | 8246
grams/deciliter (g/dL) | 14.59 (1.702) | 14 (1.909)
Statistical Analysis 1: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio (OR) = 1.050 — Odds Ratio for selection of Prasugrel for participants who had pre-procedure hemoglobin evaluation vs no hemoglobin evaluation

9. Primary Outcome: Factors Associated With Initial ADP Receptor Inhibitor Selection at Enrollment: Duke Coronary Artery Disease (CAD) Index
Description: The Duke CAD Index is a validated composite measure of angiographic burden, which assigns prognostic weights 1 through 100. Higher scores indicate greater angiographic burden and are associated with poorer prognosis.
Time Frame: Day 0 (study enrollment)
Population: All enrolled participants who had Duke CAD Index completed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prasugrel | Other
Number analyzed (Participants) | 3101 | 8923
units on a scale | 40.36 (14.43) | 41.87 (16.01)
Statistical Analysis 1: Comparison: Prasugrel; Test type: Superiority or Other; Odds Ratio (OR) = 1.005 — Odds Ratio for selection of Prasugrel for participants with Duke CAD Index vs no Duke CAD Index

ADVERSE EVENTS:
Description: Per protocol, this study only required the collection and further evaluation of non-endpoint serious adverse events (SAEs) in prasugrel-treated participants. SAE collection began after the participant signed informed consent until 7 days after last dose of prasugrel.
Arm/Group | Prasugrel
Serious Adverse Events (participants affected / at risk) | 865/3123
Other Adverse Events (participants affected / at risk) | 0/3123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Prasugrel (N=3123)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 26 (26)
Angina pectoris (Cardiac disorders) | 23 (23)
Angina unstable (Cardiac disorders) | 24 (25)
Arrhythmia (Cardiac disorders) | 7 (7)
Arteriosclerosis coronary artery (Cardiac disorders) | 25 (25)
Atrial fibrillation (Cardiac disorders) | 9 (11)
Atrial flutter (Cardiac disorders) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 7 (7)
Cardiac disorder (Cardiac disorders) | 3 (3)
Cardiac failure (Cardiac disorders) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 7 (7)
Cardiac failure congestive (Cardiac disorders) | 19 (22)
Cardiac flutter (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 6 (6)
Dressler's syndrome (Cardiac disorders) | 3 (3)
Hypertensive heart disease (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 109 (136)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 7 (8)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Amaurosis (Eye disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7)
Colitis (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 2 (2)
Gastric disorder (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (4)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (9)
Gastrointestinal inflammation (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 3 (4)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Oesophageal haemorrhage (Gastrointestinal disorders) | 2 (2)
Oesophageal rupture (Gastrointestinal disorders) | 2 (2)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (10)
Adverse drug reaction (General disorders) | 6 (6)
Arterial restenosis (General disorders) | 1 (1)
Asthenia (General disorders) | 3 (4)
Chest discomfort (General disorders) | 12 (12)
Chest pain (General disorders) | 247 (309)
Coronary artery restenosis (General disorders) | 3 (3)
Death (General disorders) | 50 (53)
Device damage (General disorders) | 1 (1)
Device dislocation (General disorders) | 1 (1)
Device failure (General disorders) | 1 (1)
Device issue (General disorders) | 1 (1)
Device malfunction (General disorders) | 2 (2)
Device occlusion (General disorders) | 6 (6)
Effusion (General disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Feeling abnormal (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Hyperthermia (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Malaise (General disorders) | 3 (4)
Non-cardiac chest pain (General disorders) | 7 (8)
Oedema (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Peripheral swelling (General disorders) | 3 (5)
Pyrexia (General disorders) | 2 (2)
Stent malfunction (General disorders) | 4 (4)
Swelling (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 9 (9)
Ulcer haemorrhage (General disorders) | 7 (7)
Unevaluable event (General disorders) | 3 (3)
Vessel puncture site haemorrhage (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 8 (8)
Abscess (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 7 (7)
Cellulitis (Infections and infestations) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 1 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 3 (3)
Device related infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Escherichia infection (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Groin infection (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (2)
Infection (Infections and infestations) | 4 (4)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Kidney infection (Infections and infestations) | 4 (4)
Localised infection (Infections and infestations) | 2 (2)
Meningitis (Infections and infestations) | 1 (1)
Orchitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 21 (22)
Sepsis (Infections and infestations) | 3 (3)
Septic shock (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 10 (10)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 6 (6)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 4 (4)
Overdose (Injury, poisoning and procedural complications) | 2 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 5 (5)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 4 (5)
Angiogram (Investigations) | 1 (1)
Aspiration pleural cavity (Investigations) | 1 (1)
Barium enema (Investigations) | 1 (1)
Biopsy lung (Investigations) | 1 (1)
Blood glucose abnormal (Investigations) | 2 (3)
Blood glucose decreased (Investigations) | 2 (2)
Blood glucose fluctuation (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 3 (3)
Blood potassium decreased (Investigations) | 2 (2)
Blood potassium increased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 4 (4)
Blood pressure increased (Investigations) | 6 (6)
Blood triglycerides increased (Investigations) | 1 (1)
Blood urine present (Investigations) | 2 (2)
Cardiac stress test (Investigations) | 2 (2)
Catheterisation cardiac (Investigations) | 81 (87)
Colonoscopy (Investigations) | 3 (3)
Computerised tomogram (Investigations) | 1 (1)
Electrocardiogram (Investigations) | 1 (1)
Electrocardiogram abnormal (Investigations) | 3 (3)
Endoscopy (Investigations) | 1 (1)
Enzyme level increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3)
Haemoglobin increased (Investigations) | 1 (1)
Heart rate abnormal (Investigations) | 1 (1)
Heart rate decreased (Investigations) | 2 (2)
Heart rate increased (Investigations) | 4 (4)
Heart rate irregular (Investigations) | 2 (2)
Imaging procedure (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Oesophagogastroduodenoscopy (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 9 (9)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (5)
Diabetic complication (Metabolism and nutrition disorders) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 3 (3)
Gout (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (10)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 4 (4)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain injury (Nervous system disorders) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 17 (22)
Coma (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 3 (3)
Dementia (Nervous system disorders) | 1 (1)
Diabetic coma (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 20 (21)
Dyskinesia (Nervous system disorders) | 2 (2)
Embolic cerebral infarction (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 6 (6)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 8 (8)
Migraine (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 12 (12)
Thrombotic stroke (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 5 (5)
Unresponsive to stimuli (Nervous system disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (7)
Confusional state (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Fear (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 2 (2)
Mental disorder (Psychiatric disorders) | 1 (1)
Neurosis (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 7 (7)
Renal failure (Renal and urinary disorders) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1/672 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1/672 (1)
Prostatic haemorrhage (Reproductive system and breast disorders) | 1/2451 (1)
Testicular swelling (Reproductive system and breast disorders) | 1/2451 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2/672 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 (59)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Angioplasty (Surgical and medical procedures) | 5 (5)
Antibiotic therapy (Surgical and medical procedures) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 1 (1)
Bladder irrigation (Surgical and medical procedures) | 1 (2)
Cardiac ablation (Surgical and medical procedures) | 2 (2)
Cardiac operation (Surgical and medical procedures) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 3 (3)
Cholecystostomy (Surgical and medical procedures) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 32 (32)
Coronary artery bypass (Surgical and medical procedures) | 9 (9)
Coronary revascularisation (Surgical and medical procedures) | 2 (2)
Dialysis (Surgical and medical procedures) | 2 (2)
Emergency care (Surgical and medical procedures) | 1 (1)
Exploratory operation (Surgical and medical procedures) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 9 (9)
Implantable defibrillator insertion (Surgical and medical procedures) | 4 (4)
Medical device removal (Surgical and medical procedures) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1)
Stent placement (Surgical and medical procedures) | 24 (24)
Surgery (Surgical and medical procedures) | 2 (3)
Therapy change (Surgical and medical procedures) | 1 (2)
Transfusion (Surgical and medical procedures) | 1 (1)
Vascular cauterisation (Surgical and medical procedures) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 39 (39)
Hypertension (Vascular disorders) | 10 (11)
Hypotension (Vascular disorders) | 6 (6)
Neurogenic shock (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 2 (2)
Shock (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 7 (7)
Vasculitis (Vascular disorders) | 1 (1)
Venous occlusion (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days